CLINICAL TRIAL: NCT02078960
Title: An Open-Label, Single-Group Clinical Study to Evaluate the Pharmacokinetics, Safety,and Efficacy of Omacetaxine Mepesuccinate Given Subcutaneously as a Fixed Dose inPatients With Chronic Phase or Accelerated Phase Chronic Myeloid Leukemia Who Have Failed 2 or More Tyrosine Kinase Inhibitor Therapies
Brief Title: A Study to Evaluate the Pharmacokinetics, Safety,and Efficacy of Omacetaxine Given Subcutaneously as a Fixed Dose in Patients With Chronic Phase (CP) or Accelerated Phase (AP) Chronic Myeloid Leukemia (CML) (Referred to as the SYNSINCT Study)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Inability to accrue additional sites and enroll an adequate number of subjects.
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C41443/2057; 2013-005320-42 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-05 (Estimated); Results first posted 2019-01-14 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Phase; Accelerated Phase; CML; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Omacetaxine mepesuccinate. (Experimental): The study will consist of up to a 7-day screening period, and treatment for up to 12 months, in Phase 1 and Phase 2 portions, depending on response and tolerability. Patients will also have an end-of-treatment follow-up visit approximately 28 days after the last dose of omacetaxine. Each patient will be monitored for progression and survival for at least 1 year after their last dose of omacetaxine, death, or lost to follow-up, whichever comes first, regardless of patients receiving other anticancer treatment.
  Interventions: Drug: Omacetaxine mepesuccinate

INTERVENTIONS:
Drug: Omacetaxine mepesuccinate — 3.5 mg omacetaxine mepesuccinate and 10 mg mannitol; The first dose of the day for cycle 1 will be administered at the investigational center. Subsequent doses (in prefilled syringes) may be administered on an outpatient basis after training takes place
  Other Names: C41443; SYNRIBO®

SUMMARY:
To satisfy a postmarketing requirement, the sponsor has been requested to conduct a Phase 1/Phase 2 single-group clinical study to investigate the pharmacokinetics and preliminary safety and efficacy of omacetaxine following a fixed-dose administration to patients with CP or AP CML who have failed 2 or more tyrosine kinase inhibitor (TKI) therapies.

DETAILED DESCRIPTION:
Because the trial was not feasible due to the inability to accrue additional clinical study sites and enroll an adequate number of subjects, the FDA released the sponsor from the postmarketing requirement on 13 November 2017 and the study was stopped prematurely. Therefore, the study did not progress to the Phase 2 portion.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a confirmed diagnosis of Philadelphia chromosome (Ph) positive chronic myelogenous leukemia in either CP or AP. Accelerated phase will be defined as disease having 1 of the following: ≥15% to <30% blasts in peripheral blood or bone marrow; ≥30% blasts + promyelocytes in peripheral blood or bone marrow; ≥20% basophils in peripheral blood or bone marrow; platelet count <100x109/L unrelated to therapy; or clonal evolution.
* The patient has either failed, demonstrated intolerance, or a combination of prior failure and intolerance, to prior treatments with at least 2 tyrosine kinase inhibitors (TKI's). Failure of TKI treatment may either be primary (never achieved a response) or secondary resistance (loss of response).
* TKI treatment failure will be defined as 1 of the following:

  * no CHR by 12 weeks (whether lost or never achieved)
  * no partial cytogenetic response by 24 weeks (ie, 1 to 35% Ph-positive) (whether lost or never achieved) no major cytogenetic response by 52 weeks (ie, ≤35% Ph-positive) (whether lost or never achieved)
  * progressive leukocytosis, defined as increasing white blood cell (WBC) count on at least 2 consecutive evaluations, at least 2 weeks apart and doubling from the nadir to ≥20000/μL or absolute increase in WBC by ≥50000/μL above the post-treatment nadir
* Intolerance to TKI therapy will be defined as 1 of the following:

  * grade 3 to 4 nonhematologic toxicity that does not resolve with adequate intervention
  * grade 4 hematologic toxicity lasting more than 7 days, or a documented inability to sustain the TKI therapy because of recurrent grade 3 or 4 hematologic toxicity with re-initiation of the same therapy
  * any grade 2 or greater toxicity that is unacceptable to the patient
* Patients must have completed all previous anticancer therapy for at least 2 weeks prior to the first planned dose of omacetaxine, except as noted below, and must have fully recovered from side effects of a previous therapy.
* In patients with rapidly proliferating disease, hydroxyurea may be administered before study entry, if clinically indicated, to control disease. In such cases, complete hematologic response (CHR) must be sustained for at least 4 weeks for accelerated CML, and at least 8 weeks for chronic phase CML, following the discontinuation of hydroxyurea, to be considered as a CHR.
* Patients may receive anagrelide for up to 28 days (in countries where the product is registered). Leukapheresis is allowed up to 24 hours prior to the first treatment cycle with omacetaxine.
* Patients must have adequate hepatic and renal function as evidenced by bilirubin 2.0 times the upper limit of the normal range (ULN) or lower, alanine aminotransferase (ALT) and asparate aminotransferase (AST) 3 times the ULN or lower, serum creatinine 1.5 times the ULN or lower. Patients with nonclinically significant elevations of bilirubin up to 5.0 g/dL (85500 μmol/L) due to known or suspected Gilbert's disease are eligible; this must be documented on the medical history page of the case report form (CRF).
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients are men or women at least 18 years of age.
* Patients must be able and willing to provide written informed consent prior to any study related procedure.
* The patient must take precautions to not become pregnant or produce offspring. Women must be of non-childbearing potential (surgically sterile or postmenopausal for at least 12 months, confirmed by follicle-stimulating hormone [FSH] >40 IU/L) or agree to use a medically accepted method of contraception for the duration of the study and 90 days after treatment. Men must be surgically sterile or agree to use a medically accepted method of contraception for the duration of the study and 90 days after treatment. Acceptable methods of contraception include abstinence, barrier method with spermicide (excluding cervical cap and sponge), intrauterine device (IUD), or steroidal contraceptive (oral, transdermal, implanted, and injected) in conjunction with a barrier method.

  * Other criteria may apply, please contact the investigator for additional information

Exclusion Criteria:

* The patient has New York Heart Association (NYHA) class III or IV heart disease, active ischemia, or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy, uncontrolled hypertension, or congestive heart failure.
* The patient has had a myocardial infarction in the previous 12 weeks. (Prior to study entry, electrocardiogram [ECG] abnormalities at screening must be documented by the investigator as not medically relevant.)
* The patient has received radiotherapy within 30 days prior to the start of study drug, or has not recovered from the acute toxicities associated with prior approved therapies including investigational drugs.
* The patient has another concurrent illness that would preclude study conduct and assessment, including, but not limited to, another active malignancy (excluding squamous or basal cell skin cancer and in situ cervical cancer), uncontrolled medical conditions, uncontrolled and active infection (considered opportunistic, life threatening, or clinically significant), uncontrolled risk of bleeding, or uncontrolled diabetes mellitus.
* The patient underwent autologous or allogeneic stem cell transplant within 60 days prior to receiving the first dose of omacetaxine and has any evidence of ongoing graft versus host disease (GVHD), or GVHD requiring immunosuppressive therapy.
* The patient has a human leukocyte antigen (HLA)-matched donor and is eligible for allogeneic transplantation for CML treatment.
* The patient has known positive human immunodeficiency virus (HIV) or known active human t-cell lymphotropic virus (HTLV) I/II disease, whether on treatment or not.
* The patient has known active hepatitis B or C. The determination of active hepatitis B or C is left to the investigator.
* The patient has lymphoid Ph+ blast crisis or blast phase CML.
* The patient participated in another clinical investigation within 30 days of enrollment or is receiving another investigational agent.
* The patient received omacetaxine or has a history of hypersensitivity.

  * Other criteria may apply, please contact the investigator for additional information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-10-09 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (10):
- United States (6):
  - Teva Investigational Site 12545, Jacksonville, Florida
  - Teva Investigational Site 12550, Atlanta, Georgia
  - Teva Investigational Site 12543, Indianapolis, Indiana
  - Teva Investigational Site 12547, Buffalo, New York
  - Teva Investigational Site 12546, Cincinnati, Ohio
  - Teva Investigational Site 12544, Houston, Texas
- Belgium (2):
  - Teva Investigational Site 37048, Ghent
  - Teva Investigational Site 37047, Leuven
- Teva Investigational Site 35157, Pierre-Bénite, France
- Teva Investigational Site 87026, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 14 patients with chronic myeloid leukemia were screened for enrollment into this study. Of the 4 patients who were not enrolled, 2 were excluded on the basis of inclusion/exclusion criteria and 2 for "other" reasons.
Pre-assignment Details: Of the 14 patients screened, 9 patients at 3 centers in the US and 1 patient at a single centre in France met entry criteria and were considered to be eligible for enrollment into the study.
Groups:
- Cohort 1: Participants whose body surface area (BSA) is less than 1.7 m^2. All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily. Induction cycles of 14 days twice daily treatment were followed by 14 days without treatment (1 induction cycle) for as long as they adequately recover their blood counts and/or until they achieve hematologic response. [Cycle 1 was an exception since participants were not dosed a second time on Day 1, nor at all on Days 2+3 to accommodate the PK study objective.] Participants then received maintenance cycles of 7 days twice daily treatment followed by 21 days without treatment (1 maintenance cycle) for as long as they continued to benefit up to a period of 12 months following the first dose.
- Cohort 2: Participants whose body surface area (BSA) is between 1.7 m^2 to 2.0 m^2 inclusive All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily. Induction cycles of 14 days twice daily treatment were followed by 14 days without treatment (1 induction cycle) for as long as they adequately recover their blood counts and/or until they achieve hematologic response. [Cycle 1 was an exception since participants were not dosed a second time on Day 1, nor at all on Days 2+3 to accommodate the PK study objective.] Participants then received maintenance cycles of 7 days twice daily treatment followed by 21 days without treatment (1 maintenance cycle) for as long as they continued to benefit up to a period of 12 months following the first dose.
- Cohort 3: Participants whose body surface area (BSA) is greater than 2.0 m^2. All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily. Induction cycles of 14 days twice daily treatment were followed by 14 days without treatment (1 induction cycle) for as long as they adequately recover their blood counts and/or until they achieve hematologic response. [Cycle 1 was an exception since participants were not dosed a second time on Day 1, nor at all on Days 2+3 to accommodate the PK study objective.] Participants then received maintenance cycles of 7 days twice daily treatment followed by 21 days without treatment (1 maintenance cycle) for as long as they continued to benefit up to a period of 12 months following the first dose.
Period: Treatment Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 2 | 4 | 4
Completed (Treatment completed) | 0 | 1 | 1
Not Completed | 2 | 3 | 3
Not completed — Other | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Disease progression - accelerated phase | 0 | 1 | 0
Not completed — Disease progression - blast phase | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1
Period: Follow-up Period
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Started | 2 | 2 | 1
Completed (Monitored for progression and survival for at least 1 year following treatment.) | 0 | 1 | 1
Not Completed | 2 | 1 | 0
Not completed — Death | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Total
Number analyzed (Participants) | 2 | 4 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 1 | 5
  >=65 years | 1 | 1 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (9.19) | 46.3 (22.87) | 68.3 (17.31) | 59.1 (20.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 2 | 3 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 1 | 2 | 4 | 7
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 2 | 4 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Weight [Mean (Standard Deviation); unit: kg] | 55.1 (7.78) | 73.7 (4.58) | 105.3 (18.34) | 82.6 (23.63)
Height [Mean (Standard Deviation); unit: cm] | 167.0 (1.41) | 167.3 (8.02) | 169.7 (9.55) | 168.2 (7.33)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] | 1.6 (0.08) | 1.8 (0.09) | 2.2 (0.25) | 2.0 (0.30)
Phase of Chronic Myeloid Leukemia (CML) at Study Entry [Count of Participants; unit: Participants] — CP: patients typically have less than 10% blasts in their blood or bone marrow samples. Patients usually have fairly mild symptoms and usually respond to standard treatments.
  AP: patients have >=1 of the following:
  * Blood samples have 15% or more, but fewer than 30% blasts
  * Basophils make up 20% or more of the blood
  * Blasts and promyelocytes combined make up 30% or more of the blood
  * Very low platelet counts (100*1,000/mm^3 or less) that are not caused by treatment
  * New chromosome changes in the leukemia cells with the Philadelphia chromosome.
  Participants
    Chronic Phase (CP) | 2 | 3 | 4 | 9
    Accelerated Phase (AP) | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Major Response at Any Time During Treatment
Description: The Independent Data Monitoring Committee assessments are summarized. Major response for participants with chronic phase CML was a major cytogenetic response (MCyR) defined as a complete cytogenetic response with no Ph+ metaphases, or a partial cytogenetic response with up to 35% Ph+ metaphases. Note that a complete hematologic response was not considered a major response.
  Major response for participants with accelerated phase CML was a major hematologic response (MaHR) defined as a complete hematologic response or no evidence of leukemia, and/or a major cytogenic response (MCyR).
Time Frame: Day 1 up to Month 15 (longest treatment duration)
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 2 | 4 | 4
Participants | 0 | 1 | 2

2. Secondary Outcome: Longest Duration of Response At Study Termination
Description: Duration of response was defined for responders as the time interval from the first reported date of a major cytogenetic response (MCyR) or a major hematologic response (MaHR) to the earliest date of objective evidence of disease progression (ie, development of accelerated-phase CML), relapse (ie, loss of complete hematologic or major cytogenetic response), or death. Kaplan-Meier estimates for duration of response were not performed due the small enrollment population and early termination of the study. What is reported is the longest duration of response observed prior to disease progression, death, lost to follow-up or study termination.
Time Frame: Day 1 to Day 541 (longest progression/survival follow-up)
Population: Enrolled participants who had a response
Measure: Number; unit: days
Groups:
- All Enrolled Participants: All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily. Induction cycles of 14 days twice daily treatment were followed by 14 days without treatment (1 induction cycle) for as long as they adequately recover their blood counts and/or until they achieve hematologic response. [Cycle 1 was an exception since participants were not dosed a second time on Day 1, nor at all on Days 2+3 to accommodate the PK study objective.] Participants then received maintenance cycles of 7 days twice daily treatment followed by 21 days without treatment (1 maintenance cycle) for as long as they continued to benefit up to a period of 12 months following the first dose.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 5
days | 316

3. Secondary Outcome: Number of Participants Who Had a Molecular Response at Any Time During Treatment
Description: Molecular response was defined by the decrease in the amount of BCR-ABL (an abnormality of chromosome 22) messenger ribonucleic acid (mRNA) measured by reverse transcriptase polymerase chain reaction (RT-PCR) or by the actual percentage of BCR-ABL mRNA transcripts (ratio of BCR-ABL transcript numbers to the number of control gene transcripts).
Time Frame: Day 1 up to Month 15
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 10
Participants | 1

4. Secondary Outcome: Number of Participants Who Were Alive and Progression-Free at Study Termination
Description: Progression-free survival was defined as the time interval from the date of first dose to the date of the earliest objective evidence of disease progression (ie, development of accelerated-phase CML), relapse (ie, loss of complete hematologic or major cytogenetic response), or death. Kaplan-Meier estimates for time for progression-free survival were not performed due the small enrollment population and early termination of the study. What is reported is the number of participants who were alive and progression-free at the time of study termination.
Time Frame: Day 1 to Day 541 (longest progression/survival follow-up)
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 10
Participants | 4

5. Secondary Outcome: Number of Participants Who Were Alive at Study Termination
Description: Overall survival was defined as the time interval from the date of the first dose to the date of death from any cause. Kaplan-Meier time estimates for overall survival were not performed due to the small enrollment population and early termination of the study. What is reported is the number of participants who were alive at the time of study termination.
Time Frame: Day 1 to Day 541 (longest progression/survival follow-up)
Population: Enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 10
Participants | 7

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Omacetaxine
Description: Maximum observed plasma drug concentration (Cmax) by inspection (without interpolation). Nominal PK sampling times were used.
Time Frame: Cycle 1 - Day 1 (predose, 15, 30, 45 minutes, 1, 2, 4, 8, 24, 48, 72 hours post-dose) Day 10 (predose, 2 samples postdose), Day 13 (predose) Cycles 2+3 - Day 1 (2 samples postdose), Days 10 and 17 (1 sample predose)
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Total Omacetaxine: All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily. Induction cycles of 14 days twice daily treatment were followed by 14 days without treatment (1 induction cycle) for as long as they adequately recover their blood counts and/or until they achieve hematologic response. [Cycle 1 was an exception since participants were not dosed a second time on Day 1, nor at all on Days 2+3 to accommodate the PK study objective.] Participants then received maintenance cycles of 7 days twice daily treatment followed by 21 days without treatment (1 maintenance cycle) for as long as they continued to benefit up to a period of 12 months following the first dose.
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
ng/mL | 23.88 (13.32)

7. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Cmax) for Omacetaxine
Description: Time to maximum observed plasma drug concentration (Cmax) by inspection (without interpolation). Nominal PK sampling times were used.
Time Frame: as for outcome 6
Population: PK analysis set
Measure: Median (Full Range); unit: hour
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
hour | 0.25 [0.25 to 1.0]

8. Secondary Outcome: Area Under the Drug Concentration by Time Curve From Time 0 to the Time of the Last Measurable Drug Concentration (AUC0-t) for Omacetaxine
Description: Nominal PK sampling times were used.
Time Frame: as for outcome 6
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
ng*hr/mL | 150.2 (55.8)

9. Secondary Outcome: Area Under the Drug Concentration by Time Curve From Time 0 to Infinity (AUC0-inf) for Omacetaxine
Description: Nominal PK sampling times were used.
Time Frame: as for outcome 6
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
ng*hr/mL | 154.8 (60.8)

10. Secondary Outcome: Terminal Elimination Half-Life (t1/2) for Omacetaxine
Description: Nominal PK sampling times were used.
Time Frame: as for outcome 6
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
hour | 13.3 (1.6)

11. Secondary Outcome: Total Oral Clearance (CL/F) for Omacetaxine
Description: Nominal PK sampling times were used.
Time Frame: as for outcome 6
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
L/hour | 18.1 (6.1)

12. Secondary Outcome: Apparent Volume of Distribution (V/F) for Omacetaxine
Description: Nominal PK sampling times were used.
Time Frame: as for outcome 6
Population: PK analysis set
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Total Omacetaxine
Number analyzed (Participants) | 10
L | 344.9 (117.0)

13. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product, regardless of whether it has a causal relationship with this treatment. A treatment-emergent adverse event (TEAE) is an AE that that began or worsened after treatment with study drug. Severity rating of 3=Severe or medically significant but not immediately life-threatening 4=Life-threatening consequences and 5=Death. Relation to study drug is determined by the investigator. A serious adverse event (SAE) includes death, a life-threatening AE, hospitalization, persistent or significant disability or incapacity, a congenital anomaly/birth defect, or any important medical event requiring immediate intervention to prevent one of the outcomes above.
Time Frame: Day 1 up to Month 15
Population: Safety Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3
Number analyzed (Participants) | 2 | 4 | 4
Participants
  Any TEAE | 2 | 4 | 4
  TEAE of Severity Grade 3 | 0 | 3 | 0
  TEAE of Severity Grade 4 | 1 | 1 | 3
  TEAE of Severity Grade 5 | 1 | 0 | 1
  Treatment-related TEAE | 2 | 4 | 4
  Deaths | 2 | 0 | 1
  Serious AE | 2 | 2 | 4
  Withdrawn from treatment due to a TEAE | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 1 up to Month 15
Groups:
- COHORT 1: Participants whose body surface area (BSA) is less than 1.7 m^2. All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily.
- COHORT 2: Participants whose body surface area (BSA) is between 1.7 m^2 to 2.0 m^2 inclusive All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily.
- COHORT 3: Participants whose body surface area (BSA) is greater than 2.0 m^2. All participants were given a fixed dose of 2.5 mg omacetaxine by subcutaneous injection twice daily.
Arm/Group | COHORT 1 | COHORT 2 | COHORT 3
All-Cause Mortality (participants affected / at risk) | 2/2 | 0/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 2/2 | 2/4 | 4/4
Other Adverse Events (participants affected / at risk) | 2/2 | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=2) | COHORT 2 (N=4) | COHORT 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (2)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COHORT 1 (N=2) | COHORT 2 (N=4) | COHORT 3 (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 (5) | 1 (1) | 2 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hypofibrinogenaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (10)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (7) | 1 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (7) | 1 (9)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (7) | 2 (10)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (5) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 1 (5) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (2) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Legionella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urethritis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Small sample size made it not possible to make meaningful comparisons between cohorts.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.

DOCUMENTS (2):
  • Study Protocol (2015-04-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT02078960/Prot_001.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT02078960/SAP_000.pdf